CLINICAL TRIAL: NCT03601858
Title: Descriptive Epidemiology of a Specialized Consultation on Attention Deficit Hyperactivity Disorder in Adults at the Strasbourg University Hospital, and Evolution Analysis at One Year
Brief Title: Descriptive Epidemiology of a Specialized Consultation on ADHD in Adults at the Strasbourg University Hospital
Acronym: Stras-TDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7083
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Attention Deficit and Hyperactivity Disorder
Keywords: Attention deficit; hyperactivity disorder; Adult; Epidemiology; Evolution; treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to carry out a descriptive study of the clinical and demographic characteristics of patients having consulted for a specialized opinion about ADHD in adults of the psychiatric service of the Strasbourg University Hospital.

The characteristics of patients were collected during the first consultation, by the psychiatrist, and analyzed retrospectively.

The secondary objective is to evaluate the evolution at one year in terms of follow-up, maintenance under medical treatment and perceived effects of it.

The patients who had a prescription for pharmacological treatment of ADHD were contacted between 9 and 15 months after the first consultation and responded to a questionnaire assessing the evolution.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Having a specialized consultation about ADHD in adults in the psychiatric service of the Strasbourg University Hospital
* Agree with the use of medical files from the consultation for medical research

Exclusion Criteria:

* Disgree with the use of medical files from the consultation for medical research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient Having a specialized consultation about ADHD in adults in the psychiatric service of the Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Hyperactivity Disorder | Between 9 and 15 months after the first consultation, contact of patients and collection of data for the evolution at one year analyze
  Measuring from the medical files of patients and questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie II, Strasbourg, France